CLINICAL TRIAL: NCT04676243
Title: Randomized Study in Newly Diagnosed AML With FLT3-ITD Comparing Daunorubicin/ Cytarabine or Idarubicin/Cytarabine and Quizartinib to Physician's Choice
Brief Title: Daunorubicin or Idarubicin With Cytarabine Plus Quizartinib vs Physician's Choice in Newly Diagnosed FLT3-ITD+ AML
Acronym: Q-SOC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study turned out no longer feasible
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Richard F Schlenk, Assistant medical director, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HeLeNe 20-04
Record Dates: First submitted 2020-12-09; First posted 2020-12-19 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML newly diagnosed; Quizartinib added to SOC; FLT3-ITD positivity
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib

STUDY DESIGN:
Intervention Model Description: multicenter, randomized phase in patients with FLT3-ITD positive AML comparing quizartinib in combination with SOC chemotherapy versus treatment according to physician's choice (PhC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quizartinib plus standard of care (SOC) (Experimental): Daunorubicin/ Cytarabine or Idarubicin/Cytarabine and Quizartinib
  Interventions: Drug: Quizartinib; Drug: Standard of Care Chemotherapy
- Physician's choice (Active Comparator): Physician's choice (usually Daunorubicin/ Cytarabine or Idarubicin/Cytarabine and Midostaurin)
  Interventions: Drug: Treatment according to Physician's Choice

INTERVENTIONS:
Drug: Quizartinib — 20 mg coated tablets, orally administered
  Other Names: Drug Code:AC220
  Arms: Quizartinib plus standard of care (SOC)
Drug: Treatment according to Physician's Choice — Usually daunorubicin/ cytarabine or idarubicin/Cytarabine plus FLT3 inhibitor (usually midostaurin)
  Other Names: PhC
  Arms: Physician's choice
Drug: Standard of Care Chemotherapy — Daunorubicin/ Cytarabine or Idarubicin/Cytarabine
  Other Names: SOC
  Arms: Quizartinib plus standard of care (SOC)

SUMMARY:
The orally administered second-generation bis-aryl urea tyrosine kinase inhibitor quizartinib is very specific for FLT3, has a high capacity for sustained FLT3-inhibition and an acceptable toxicity profile. Furthermore, single agent quizartinib doubled the response rate as compared to standard of care in a randomized study in r/r-AML. Combination therapy of quizartinib with intensive standard induction chemotherapy has been shown to be safe and moreover, single agent quizartinib maintenance therapy is feasible even after allogeneic HCT.

The efficacy of quizartinib in combination with intensive induction and post-remission therapy including allogeneic HCT and single agent quizartinib as maintenance therapy is evaluated by this protocol. This approach is compared in a randomized manner to the current standard of care.

DETAILED DESCRIPTION:
This is a multicenter, upfront randomized phase III trial of patients with FLT3-ITD positive AML comparing quizartinib in combination with SOC chemotherapy versus treatment according to physician's choice (PhC). Efficacy is assessed by comparing EFS between the quizartinib and the PhC arm of the study.

Primary objective To improve modified event-free survival (mEFS) with Quizartinib added to induction and consolidation therapy followed by single agent maintenance therapy compared to physician's choice (PhC)

Secondary objectives To improve overall survival (OS) with Quizartinib added to conventional therapy compared to physician's choice; To improve remission (including CR/CRi/CRh) rate with Quizartinib added to conventional therapy compared to physician's choice To reduce measurable residual disease (MRD) with Quizartinib added to conventional therapy compared to physician's choice after induction (MRDind), consolidation (MRDcons), before allogeneic hematopoietic cell transplantation (MRDpre-HCT ) and maintenance (MRDmaintenance) therapy Assessment of patient reported outcomes (PRO) after induction, consolidation and maintenance therapy and after two years Evaluation of safety based on duration of neutropenia and leukopenia, incidence of infection, duration of initial hospitalization and number of transfusions (e.g. packed red blood cells and platelets) Cost-effectiveness analysis of the two different treatment schedules from health care payer´s perspective.

Budget impact analysis of introducing effective treatment schedule(s) in everyday clinical practice.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of untreated acute myeloid leukemia (AML) according to the WHO 2016 definition
* Positive for FLT3-ITD (defined as a ratio of mutant to wild-type alleles of at least 0.05; measured within 4 weeks before randomization)
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis before randomization (≤7 days) *
* Age ≥18 years, no upper age limit
* ECOG PS ≤2. (Eastern Cooperative Oncology Group performance status)
* Adequate renal function defined as creatinine clearance >50 mL/min (calculated using the standard method of the local institution)
* Considered eligible to receive intensive chemotherapy as per investigator judgment
* No contraindications for FLT3-inhibitor therapy
* No severe organ function abnormalities
* Not included in other first-line trials
* Non-pregnant and non-nursing women
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 48 hours prior to randomization. ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
* WOCBP must agree to avoid getting pregnant while on therapy: WOCBP must either commit to continued abstinence from heterosexual intercourse or begin and adhere to one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy) during study and 6 months after end of study/treatment.**
* Men must use a latex condom during any sexual contact with WOCBP, even if they have undergone a successful vasectomy and must agree to avoid to father a child during study and 6 months after end of study/treatment
* Signed written informed consent
* Ability of patient to understand character and consequences of the clinical trial
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

  * In case hyperleukocytosis is not controllable with hydroxyurea, treatment with e.g. cytarabine should be discussed in Germany with the principal investigator and in Spain with the PETHEMA trials office or for patients of both countries with the medical coordinator.

    * A high follicle-stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy at investigator's discretion.

Exclusion Criteria

* AML with PML-RARA or BCR-ABL1
* Patients with known active central nervous system (CNS) leukemia (assessed clinically).
* Isolated extramedullary manifestation of AML
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy for more than one year and are considered by their physician to be at less than 30% risk of relapse within one year.
* Prior treatment for AML, except for the following allowances:

  * Leukapheresis;
  * Treatment for hyperleukocytosis with hydroxyurea;
  * Cranial radiotherapy for central nervous system (CNS) leukostasis;
  * Prophylactic intrathecal chemotherapy;
  * Growth factor/cytokine support;
* Uncontrolled or significant cardiovascular disease, including any of the following:

  * History of heart failure NYHA class 3 or 4
  * Left ventricular ejection fraction (LVEF) ≤40% by echocardiogram (ECHO)
  * History of uncontrolled angina pectoris or myocardial infarction within 12 months prior to screening
  * History of second (Mobitz II) or third degree heart block or any cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Inadequate liver function at screening: ALT and AST ≥2.5 x ULN), total bilirubin ≥1.5 x ULN; Alkaline phosphatase ≥2.5 x ULN. Known liver cirrhosis or history of Sinusoidal Obstruction Syndrome (SOS)
* Known positivity for HIV, active HBV, HCV or hepatitis A infection (active hepatitis HBV defined by HBsAg positivity, active HCV defined by positive virus load)
* Uncontrolled active infection
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy
* Any one of the following ongoing or present in the previous 6 months: congenital long QT syndrome, Torsades de Pointes, arrhythmias (including sustained ventricular tachyarrhythmia), right or left bundle branch block and bifascicular block, unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism; as well as bradycardia defined as <50 bpms
* QTc interval at screening >450 msec using the Fredericia correction (QTcF).
* Patients known to be refractory to platelet or packed red cell transfusions as per institutional guidelines, or who are known to refuse or who are likely to refuse blood product support.
* Severe neurologic or psychiatric disorder interfering with ability of giving informed consent
* Known or suspected active alcohol or drug abuse
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as informing the family physician about study participation.
* Pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Prior treatment with quizartinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Modified Event-free survival (mEFS) | through study completion (up to 4 years), from randomization until occurence of event a) b) or c) on individial patients' basis
  mEFS is defined as the time from randomization until one of the following events, whichever occurs first: a) failure to obtain complete remission (CR) or complete remission with incomplete hematological recovery (CRi) or CR with partial recovery of peripheral blood counts (CRh) after induction therapy including one or two induction treatment cycles limited to an observational period of maximally 100 days, b) relapse from CR/CRi/CRh or c) death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion (up to 4 years), frome randomization until death from any cause
  OS is defined as the time from randomization to time of death from any cause. Patients without event are censored on the last date of follow-up.
Composite remission | End of induction therapy, between 4 and 12 weeks
  Composite remission is defined as the proportion of patients experiencing a CR/CRi/CRh after induction therapy.
Measurable residual disease (MRD) | End of induction thearpy (28-84 days from randomization), End of consolidation therapy (140-222 days from randomization), End of maintenance therapy (140-1,120 days from randomization)
  MRD after induction (MRDind), consolidation (MRDcons), and maintenance (MRDmaintenance) therapy, MRD is assessed by flow cytometry according to European Leukemia Net recommendations (Döhner et al, Blood 2017;129(4):424-447.)

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, Prof Dr, Principal Investigator — NCT Trial Center, University Heidelberg

IPD SHARING:
Plan to Share IPD: No